CLINICAL TRIAL: NCT02433756
Title: Responders and Quadripolar LV Lead in CRT
Acronym: ResQ CRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Santa Croce-Carle Cuneo (Other)
Responsible Party: Principal Investigator, Antonello Vado, MD, Ospedale Santa Croce-Carle Cuneo
Other Study IDs: 001
Record Dates: First submitted 2015-04-22; First posted 2015-05-05 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months

INTERVENTIONS:
Device: CRTD

SUMMARY:
The purpose of this study is to observe the evolution of the CRTD system with left quadripolar lead, in terms of electrical parameters in all pacing configurations and to evaluate the impact on the clinical outcome.

DETAILED DESCRIPTION:
Cardiac resynchronization therapy (CRT) is limited by a high proportion of non-responders.

Pacing activation from proximal area with a left quadripolar lead might improve the depolarization pattern.

To explore the effect of CRT pacing on cardiac activity, the investigators will enroll approximately 180 patients who already underwent CRT-D implantation with a quadripolar LV lead.

After implant, as clinical practice, the device will be programmed with distal LV pacing configuration, after 6 months in patient non-responders to CRT therapy the pacing configuration will be changed (proximal configuration).

After 12 months in patients non-responders will be changed the pacing configuration again, choosing, if it is possible, a multi point pacing (pacing activation from multiple separated left ventricular (LV) sites).

ELIGIBILITY:
Inclusion Criteria:

* Be in NYHA II, III or IV functional class with approved standard indication by ESC/EHRA Guidelines
* Successful quadripolar LV lead implant

Exclusion Criteria:

* Less than 18 years of age
* Epicardial Lead
* Life expectancy < 12 months
* Pregnant or are planning to become pregnant during the duration of the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients presenting improving in Heart Failure Clinical Composite and reverse remodeling after 6 months | 6-Months
Percentage of patients presenting improving in Heart Failure Clinical Composite and reverse remodeling after 12 months | 12-Months

SECONDARY OUTCOMES:
Percentage of patients presenting improving in Heart Failure Clinical Composite and reverse remodeling after 18 months | 18 months

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Ciriè Hospital, Cirié
  - S.Croce e Carle Hospital, Cuneo
  - Maria Vittoria Hospital, Torino